CLINICAL TRIAL: NCT04654741
Title: The Rate of Embryo Euploidy in Women Treated With Progestin-primed Ovarian Stimulation Versus Conventional Ovarian Stimulation: a Randomized Controlled Trial
Brief Title: The Rate of Embryo Euploidy in Progestin-primed Ovarian Stimulation Cycles
Acronym: PPOS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Casa di Cura Privata Villa Mafalda (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4/2018
Record Dates: First submitted 2020-11-22; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: IVF; Infertility
Keywords: PGT-A; IVF; ICSI; Blastocyst; GnRH antagonist; Progestin
MeSH Terms: conditions — Infertility | interventions — Medroxyprogesterone Acetate; ganirelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Progestin Primed ovarian stimulation Group (Experimental): progestin 10 mg daily during ovarian stimulation
  Interventions: Drug: Medroxyprogesterone Acetate
- GnRH antagonist (Active Comparator): GnRH antagonist 0.25 mg daily during ovarian stimulation
  Interventions: Drug: Ganirelix Acetate

INTERVENTIONS:
Drug: Medroxyprogesterone Acetate — 1 pill per day
  Other Names: Farlutal
  Arms: Progestin Primed ovarian stimulation Group
Drug: Ganirelix Acetate — 1 injection per day
  Other Names: Orgalutran
  Arms: GnRH antagonist

SUMMARY:
The main objective of this non-inferiority randomized controlled trial is to assess the rate of blastocyst euploidy and the number of euploid blastocysts in women undergoing IVF/ICSI and treated with PPOS versus conventional ovarian stimulation based on the use of GnRH antagonist The hypothesis is that PPOS is associated with a rate of blastocyst euploidy similar to what found with the conventional ovarian stimulation. In other words, the number of euploid blastocysts that can be obtained with the PPOS strategy is expected to be the same obtained with conventional ovarian stimulation.

Moreover we expect to find non significant differences in all intermediate outcome of the IVF cycles, such as in the rate of premature LH surge, in the rate of patients with elevation of Progesterone on the triggering day, in FSH consumption and length of stimulation, in the rate of poor response and hyperresponse, in number of retrieved and mature oocytes, in fertilization and blastulation rate, in the number of available blastocysts and in the morphological quality of blastocysts

DETAILED DESCRIPTION:
The study proposed is a non-inferiority randomized controlled trial Only patients undergoing PGT-A could be included. PGT-A will be proposed to couples for reasons of advanced maternal age, recurrent miscarriage, repeated implantation failure, or severe male infertility, as well as to all good-prognosis patients who desire information regarding the health status of their embryos.

396 patients will be included in this study (198 per arm). After randomization, patients will be treated according to the PPOS or conventional ovarian stimulation strategy. For all patients the ICSI and PGT-A will be applied and the intermediate and definitive outcomes of the ART cycles will be recorded.

Ovarian Stimulation Controlled ovarian stimulation will start on the second day of the menstrual cycle, with an initial dose of recombinant follicle stimulating hormone (rFSH) (chosen according to age, antral follicle count or serum AMH and body mass index,BMI) In addition to the gonadotrophin, participants will receive progestins (MPA) in the PPOS or GnRH antagonists in the conventional ovarian stimulation. Ovarian stimulation will culminate with the oocyte retrieval procedure.

Oocyte Insemination, Embryo Culture, and Biopsy. All biologic procedures will be performed as already described. Only oocytes with the first polar body extruded (metaphase II) will be treated with the use of ICSI immediately after the denudation procedure. Finally, injected oocytes will be moved to single drops of cleavage medium. Depending on the embryo's development, the blastocyst stage can be reached on day 5, 6, or 7. On the day of biopsy, 5-10 trophectoderm cells will be gently aspirated into the biopsy pipette followed by a laser-assisted removal from the rest of the blastocyst. Briefly, trophectoderm cell samples and negative controls will be processed according to the Illumina protocol.

ELIGIBILITY:
Inclusion Criteria:

* advanced maternal age,
* recurrent miscarriage,
* repeated implantation failure,
* severe male infertility,
* patients who desire information regarding the health status of their embryos.

Exclusion Criteria:

* Ovarian cyst,
* previous surgery,
* abnormal karyotype,
* genetic or systematic disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 396 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
blastocyst euploidy | From the date of randomization up to the assessment of blastocyst euploidy (up to 20 weeks)
  the rate of blastocyst euploidy

SECONDARY OUTCOMES:
premature lh surge | From the date of randomization up to the completion of ovarian stimulation (up to 20 weeks)
  the rate of premature lh surge
oocytes | From the date of randomization up to the completion of ovarian stimulation (up to 20 weeks)
  number of total and mature oocytes
blastocysts | From the date of randomization up to the completion of the IVF cycle (up to 20 weeks)
  number of total and good quality blastocysts

CONTACTS AND LOCATIONS:
Locations (1):
- Villa Mafalda, Roma, Italy